CLINICAL TRIAL: NCT03168217
Title: Classification of Periodontitis Revisited: A Cluster Analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Paris 7 - Denis Diderot (Other)
Responsible Party: Principal Investigator, Hélène Rangé, Clinical Professor, University Paris 7 - Denis Diderot
Other Study IDs: 1973520
Record Dates: First submitted 2017-01-17; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Periodontitis
Keywords: Periodontitis; classification; Cluster analysis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to identify phenotypic groups of patients with periodontitis by applying a cluster analysis.

DETAILED DESCRIPTION:
This is a retrospective cross-sectional study based on a prospectively maintained database of consecutive patients attending the Departement of Periodontology at the Rothschild hospital. A cluster analysis will help to distinguish clinical and microbiological profils of periodontal patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with periodontitis either aggressive or chronic

Exclusion Criteria:

* Patients who had received periodontal therapies or antimicrobial therapy within the 6 months preceding the examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective cross-sectional analysis based on a prospectively maintained database of consecutive patients attending the Department of Periodontology at the Rothschild Hospital of Paris (France)
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2003-01; Primary Completion 2010-01 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Loss (CAL) | one day
  measured in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bouchard, PhD,DDS, Study Chair — Paris Diderot University

IPD SHARING:
Plan to Share IPD: Yes
IPD Will be shared on request